CLINICAL TRIAL: NCT00567905
Title: Effect of Green Tea Extract on Type 2 Diabetes: a Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Effect of Green Tea Extract on Type 2 Diabetes
Acronym: GTT-DM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taipei Hospital, Taiwan (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Chung-Hua Hsu, Taipei Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tpe-2007-IRB-05; NSC-96-2320-13-192-001
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Green tea extract; overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight | interventions — Tea; Cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Green tea extract
  Interventions: Dietary Supplement: Green tea extract
- B (Placebo Comparator)
  Interventions: Dietary Supplement: Green tea extract

INTERVENTIONS:
Dietary Supplement: Green tea extract — main content is epigallocatechin gallate (EGCG, 58%)
  Other Names: A:GTE (500 mg) tid/day; B:Placebo (cellulose, 500 mg) tid/day

SUMMARY:
The purpose of this study is to examine the effect of green tea extract (GTE) on type 2 diabetes and to explore the relationship between GTE and related hormone peptides.

DETAILED DESCRIPTION:
Green tea is one of the most popular beverages in the world. It is believed to have beneficial effects in prevention and treatment of many diseases, one of which is anti-obesity and anti-diabetes.

The benefit effects of green tea are mainly attributed to its polyphenol content, especially the most abundant one-epigallocatechin gallate (EGCG), which might inhibit adipocyte proliferation and differentiation in vitro studies

We hypothesized that GTE would improve insulin resistance in type 2 overweight diabetes and related hormone peptides will be influenced. Thus, we conducted this randomized clinical trial to examine the effect of GTE on type 2 diabetes and to explore the relationship between GTE and related hormone peptides.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Body mass index >25 kg/mm
* Aged between 20 and 65 years
* Being Chinese

Exclusion Criteria:

* Aminotransferases aspartate or aminotransferases alanine > 80 IU/L, serum creatinine > 2.0 mg/dl,
* Prolating or pregnant women, and patients with heart failure, acute myocardiac infarct, stroke and heavy injuries, and
* Any other conditions not suitable for trial as evaluated by the physician.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Homeostasis model assessment for insulin resistance (HOMA-IR) was used as the major outcome measurement. | 16 weeks

SECONDARY OUTCOMES:
HbA1C, blood sugar, creatinine, aminotransferases aspartate, aminotransferases alanine, uric acid, and plasma lipoproteins (triglyceride, cholesterol, cholesterol-HDL (HDL) and cholesterol-LDL (LDL)) cholesterol; BMI,WC---. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hua Hsu, MD; PhD, Study Chair — Branch of Chinese Medicine, Taipei City Hospital
Locations (2):
- Taiwan (2):
  - Branch of Chinese Medicine, Taipei City Hospital, Taipei
  - Branch of Chinese Medicine, Taipei

REFERENCES:
- [Background] Kao YH, Chang HH, Lee MJ, Chen CL. Tea, obesity, and diabetes. Mol Nutr Food Res. 2006 Feb;50(2):188-210. doi: 10.1002/mnfr.200500109. PMID 16416476
- [Derived] Hsu CH, Liao YL, Lin SC, Tsai TH, Huang CJ, Chou P. Does supplementation with green tea extract improve insulin resistance in obese type 2 diabetics? A randomized, double-blind, and placebo-controlled clinical trial. Altern Med Rev. 2011 Jun;16(2):157-63. PMID 21649457